CLINICAL TRIAL: NCT05231434
Title: Influence of Hydration and Functional Capacity on the Recovery of Nonlinear Heart Rate Dynamics in Healthy Individuals: Crossover Clinical Trial
Brief Title: Influence of Hydration and Functional Aerobic Capacity on the Nonlinear Dynamics of Heart Rate in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Luiz Carlos Marques Vanderlei, Principal Investigator, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 38152620.5.0000.5402
Record Dates: First submitted 2022-01-05; First posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Healthy
Keywords: exercise; hydration; non-linear dynamic; Autonomic nervous system
MeSH Terms: conditions — Motor Activity | interventions — Water; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control protocol (Active Comparator): The control protocol will consist of an initial 10 minutes of rest, followed by 90 minutes of aerobic activity and 60 minutes of the final recovery. Hydration will not be allowed throughout the protocol
  Interventions: Other: aerobic activity
- Hydration protocol (Experimental): The control protocol will consist of an initial 10 minutes of rest, followed by 90 minutes of aerobic activity and 60 minutes of the final recovery. In this protocol, volunteers will be hydrated with mineral water from the 15th minute of exercise until the end of recovery
  Interventions: Other: water; Other: aerobic activity

INTERVENTIONS:
Other: water — hydration with mineral water in 10 equal portions, administered at regular intervals from the 15th minute of exercise until the end of the recovery period.
  Arms: Hydration protocol
Other: aerobic activity — aerobic activity

SUMMARY:
The objective of this study is to analyze the influence of hydration and functional aerobic capacity in young and healthy individuals on non-linear heart rate dynamics as a technique that favor faster and more efficient recovery cardiac autonomic modulation.

ELIGIBILITY:
Inclusion Criteria:

* include healthy and male individuals, age between 18 and 30 years and physically active.

Exclusion Criteria:

* individuals who smoke and drink, those who have infections, metabolic and respiratory diseases that may interfere in the results and orthopedic problems.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-04-16 (Actual); Study Completion 2021-04-16 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | up to 3 weeks
  Will occur indirectly, using a stethoscope and an aneroid sphygmomanometer in the left arm. The indicated values will be registered in an individual form. To avoid errors in the determination of blood pressures in volunteers, a single evaluator will measure these variables throughout the experimental procedure. Data will be collected at the end of the 10 minutes of initial rest and at minutes 30, 60 and 90 during exercise on the treadmill, as well as will be collected at minutes 1, 5, 10, 20, 30, 40, 50 and 60 of recovery.
Heart Rate | up to 3 weeks
  The heart rate will be captured beat by beat using the Polar RS800CX frequency meter, equipment previously validated to capture this parameter. Data will be collected at the end of the 10 minutes of initial rest and at minutes 30, 60 and 90 during exercise on the treadmill, as well as will be collected at minutes 1, 5, 10, 20, 30, 40, 50 and 60 of recovery.
Autonomic Modulation - SD1 index | up to 3 weeks
  the data for this evaluation will be collected using a heart rate monitor that registers the heart rate beat by beat and provides information regarding the RR intervals. The SD1 index corresponds to the dispersion of points perpendicular to the line of identity of the ellipse obtained from the Poincaré plot. Expressed in milliseconds.
Autonomic Modulation - SD2 index | up to 3 weeks
  The data for this evaluation will be collected using a heart rate monitor that registers the heart rate beat by beat and provides information regarding the RR intervals. The SD2 index corresponds to the dispersion of points along the line of identity of the ellipse obtained from the Poincaré plot. Expressed in milliseconds.

CONTACTS AND LOCATIONS:
Overall Officials: thamyres rangel R barros, Principal Investigator — Universidade Estadual Júlio de Mesquita Filho
Locations (1):
- Universidade Estadual Júlio de Mesquita Filho, Presidente Prudente, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided